CLINICAL TRIAL: NCT03546803
Title: Assessment of 3M Cavilon Advanced Skin Protectant for the Prophylaxis of Radiation Dermatitis in Cancer Patients
Brief Title: 3M Cavilon Advanced Skin Protectant for the Prophylaxis of Radiation Dermatitis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ivy A. Petersen, M.D., Radiation Oncology Consultant, Mayo Clinic
Other Study IDs: 17-006813; ROR1603 (Other: Mayo Clinic)
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Head and Neck Patients; Photon or Proton Treatment with product
  Interventions: Other: 3M™ Cavilon™ Advanced Skin Protectant
- Cohort B: Hair/skin fold areas (Axilla, Groin, Perineum); Photon or Proton Treatment with product
  Interventions: Other: 3M™ Cavilon™ Advanced Skin Protectant
- Cohort C: Misc. (per Rad Onc Physician); Photon or Proton Therapy with routine skin care
  Interventions: Other: 3M™ Cavilon™ Advanced Skin Protectant

INTERVENTIONS:
Other: 3M™ Cavilon™ Advanced Skin Protectant — liquid skin protectant on skin to protect from radiation dermatitis

SUMMARY:
This study observes a liquid skin protectant that is a polymeric-cyanoacrylate solution designed to protect intact or damaged skin due to radiation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years.
* Patient has initial or recurrent disease
* Undergoing external beam radiotherapy at the Mayo Clinic Rochester campus Note: Patients who are undergoing concurrent chemotherapy are eligible
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to consent for photography of radiation field
* Available to return to Mayo Clinic in within 1 week post treatment for assessment (+/- 7 days).
* At risk for developing ≥ grade 2 dermatitis radiation as determined by treating Radiation Oncology clinician
* Biologic effective dose of >42 Gy10 as calculated using the web site EQD2.com.

Exclusion Criteria:

* Unable to provide informed consent
* Patients with active rash, pre-existing dermatitis, lupus or scleroderma within the treatment area that may make skin assessment for the study difficult
* Known history of developing an allergic reaction after using a product containing cyanoacrylate or acrylates
* Subject has a medical condition that in the opinion of the investigator should exclude him/her from participating in the study
* Subject has been enrolled in an investigational study where product was applied to the proposed study site within 30 days of the screening visit
* The skin area affected by radiation requires treatment with a concomitant medication or product (if applicable)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Radiation therapy patients
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
compare radiation dermatitis severity | 3 months (+/- 1 month) following the completion of radiation therapy
  To compare radiation dermatitis severity in irradiated skin protected by a liquid skin protectant (3M™ Cavilon™ Advanced Skin Protectant) that rapidly dries versus uncovered skin (internal control) as determined by a panel.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials